CLINICAL TRIAL: NCT06751186
Title: Effect of 'Teté Dance' on the Duration of the Lactation Session in Irritable Infants in Peru: a Randomized Controlled Trial
Brief Title: Effect of Teté Dance on Breastfeeding Duration in Irritable Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Crianzamor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202400018
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Breastfeeding Duration; Infant Feeding Practices
Keywords: Breastfeeding Duration; Irritable Infants; Maternal Support; Teté Dance Intervention; Breastfeeding Practices; Cultural Lactation Support; Infant Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teté Dance Intervention (Experimental): Participants in this group will receive guided sessions of the Teté Dance facilitated by trained individuals over a seven-day period to improve breastfeeding session duration.
  Interventions: Behavioral: Teté Dance Guided Support
- Standard Breastfeeding Support (No Intervention): Participants in this group will receive standard breastfeeding support as provided by usual care practices, without any additional interventions.

INTERVENTIONS:
Behavioral: Teté Dance Guided Support — A culturally tailored behavioral intervention combining physical activity and community engagement to support breastfeeding practices.
  Arms: Teté Dance Intervention

SUMMARY:
This study aims to evaluate the impact of a culturally adapted intervention, the Teté Dance, on the breastfeeding duration of irritable infants. Participants will be mothers of infants experiencing irritability during feeding. The study involves comparing two groups: an intervention group practicing the Teté Dance and a control group receiving standard breastfeeding support.

Researchers will assess breastfeeding session duration over a seven-day period to determine whether the Teté Dance helps extend feeding times. Participants in the intervention group will receive guided sessions from trained facilitators in a community setting, while the control group will continue with usual care.

By focusing on culturally sensitive practices, this research aims to provide a low-cost, practical solution for improving breastfeeding outcomes in resource-limited settings. Participants will be evaluated for eligibility based on specific criteria, including willingness to participate and the infant's health status. Results from this trial may contribute to global breastfeeding support strategies.

DETAILED DESCRIPTION:
This randomized controlled trial will investigate the effect of the Teté Dance, a culturally adapted maternal intervention, on breastfeeding session durations in irritable infants. Rooted in traditional Peruvian Amazonian practices, the Teté Dance integrates rhythmic maternal movements and cheerful music to create a calming environment conducive to prolonged breastfeeding.

The study will employ a parallel design with two groups: an intervention group practicing the Teté Dance and a control group receiving standard breastfeeding support. The intervention will be delivered through a combination of in-person and virtual training sessions led by trained facilitators, ensuring consistency in technique application. Mothers in the intervention group will be provided with resources, including tutorial videos and culturally tailored music playlists, to support implementation at home.

Data collection will focus on breastfeeding session durations over a seven-day period. Diaries maintained by mothers will be validated daily by blinded staff to ensure the accuracy and reliability of the recorded information. The trial will be structured to evaluate not only the immediate effects of the intervention but also its feasibility and acceptability as a culturally sensitive support strategy.

The Teté Dance aims to represent an innovative approach that leverages cultural traditions to address breastfeeding challenges in resource-limited settings. By combining traditional practices with modern support frameworks, this intervention seeks to provide a scalable and low-cost solution to improve breastfeeding outcomes globally.

Findings from this study are expected to contribute to the growing evidence supporting culturally adapted maternal interventions and may inform the development of public health policies aimed at reducing early breastfeeding cessation and its associated health risks.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 4 to 20 weeks.
* Infants identified as "demanding," meaning those with frequent irritability, restlessness, or excessive crying during breastfeeding attempts, without an underlying medical condition.
* Mothers who have completed secondary education.

Exclusion Criteria:

* Infants with significant clinical conditions.
* Infants with inadequate growth.
* Infants exclusively fed with formula.

Ages: 4 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Session Duration | 7 days from intervention start date.
  Measurement of the total duration of breastfeeding sessions recorded by participants in minutes. This measure aims to evaluate the impact of the Teté Dance intervention on breastfeeding behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Javier H Ravichagua Ashiyama, MD, Principal Investigator — Crianzamor
Locations (1):
- Crianzamor, Piura, Piura, Peru

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data on breastfeeding session durations measured at baseline and at the end of the intervention period. These data will be shared to facilitate secondary analyses and further research on culturally sensitive breastfeeding interventions. Data will be available upon reasonable request and approval by the study investigators.
Supporting Information: ICF
Time Frame: The individual participant data (IPD) and supporting information will be available starting from the date of publication of the primary research article and will remain accessible for one year. Researchers can request access during this period by contacting the study team.
Access Criteria: Access to the individual participant data (IPD) and supporting information will be granted to researchers affiliated with recognized institutions, organizations, or academic bodies. They will have access to the breastfeeding duration data collected at baseline and at the end of the intervention. To request access, researchers must submit a formal application detailing the purpose of use, supported by institutional approval. Data will be shared through a secure data-sharing platform upon agreement to a data-sharing contract that ensures confidentiality and proper data usage.

REFERENCES:
- [Background] Jiang H, Li M, Wen LM, Hu Q, Yang D, He G, Baur LA, Dibley MJ, Qian X. Effect of short message service on infant feeding practice: findings from a community-based study in Shanghai, China. JAMA Pediatr. 2014 May;168(5):471-8. doi: 10.1001/jamapediatrics.2014.58. PMID 24639004
- [Background] Britton C, McCormick FM, Renfrew MJ, Wade A, King SE. Support for breastfeeding mothers. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD001141. doi: 10.1002/14651858.CD001141.pub3. PMID 17253455
- [Background] Rollins NC, Bhandari N, Hajeebhoy N, Horton S, Lutter CK, Martines JC, Piwoz EG, Richter LM, Victora CG; Lancet Breastfeeding Series Group. Why invest, and what it will take to improve breastfeeding practices? Lancet. 2016 Jan 30;387(10017):491-504. doi: 10.1016/S0140-6736(15)01044-2. PMID 26869576
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Victora CG, Bahl R, Barros AJ, Franca GV, Horton S, Krasevec J, Murch S, Sankar MJ, Walker N, Rollins NC; Lancet Breastfeeding Series Group. Breastfeeding in the 21st century: epidemiology, mechanisms, and lifelong effect. Lancet. 2016 Jan 30;387(10017):475-90. doi: 10.1016/S0140-6736(15)01024-7. PMID 26869575
- [Background] Horta BL, Loret de Mola C, Victora CG. Long-term consequences of breastfeeding on cholesterol, obesity, systolic blood pressure and type 2 diabetes: a systematic review and meta-analysis. Acta Paediatr. 2015 Dec;104(467):30-7. doi: 10.1111/apa.13133. PMID 26192560
- See also: This link provides access to WHO's e-Library of Evidence for Nutrition Actions (eLENA), with guidelines on exclusive breastfeeding for optimal growth, development, and health in infants, along with public health strategies. — https://www.who.int/tools/elena/interventions/exclusive-breastfeeding